CLINICAL TRIAL: NCT01996150
Title: Assessing the Impact of Bleach Baths on Itch, Cutaneous Inflammation, Microbial Flora and Skin Barrier Function in Adult Atopic Dermatitis Subjects
Brief Title: Bleach Bath Treatment of Adults With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); National Eczema Association (Unknown)
Responsible Party: Principal Investigator, Lisa Beck, Professor of Medicine and Dermatology, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB/URMC- 2013; R21AR062357 (NIH)
Record Dates: First submitted 2013-11-12; First posted 2013-11-27 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; eczema; bleach bath; itch; skin barrier; staphylococcus aureus
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Pruritus; Staphylococcal Infections | interventions — Sodium Hypochlorite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dilute bleach bath (Experimental): Subjects will take a diluted bleach bath (0.005% Sodium hypochlorite) for 5-10 minutes twice a week for 12 weeks.
  Interventions: Drug: bleach bath (sodium hypochlorite)

INTERVENTIONS:
Drug: bleach bath (sodium hypochlorite) — Subjects will take diluted bleach bath (0.005% Sodium Hypochlorite) for 5-10 minutes twice a week for 12 weeks.
  Other Names: Sodium hypochlorite

SUMMARY:
This is pilot, mechanistic study to address whether bleach baths given to adult subjects with atopic dermatitis or eczema, who are colonized with the bacteria Staphylococcus aureus, will significantly alter their skin microbiome and in so doing improve their skin barrier, diminish expression of inflammatory proteins in the skin and improve itch. To answer these questions the investigators will perform a 3-month, pilot, investigator-initiated, single-center, open-label clinical study. This study will allow us to test the following hypothesis: 1) that bleach baths will normalize skin barrier function, 2) that bleach baths will diminish the local inflammatory response in the skin, and 3) that bleach baths will improve validated measures of itch (also called pruritus).

DETAILED DESCRIPTION:
Atopic Dermatitis subjects have different proportions of bacterial communities on their skin surface. Often, their skin is colonized with the pathogenic bacteria called Staphylococcus aureus. Studies have demonstrated a remarkable clinical improvement in Atopic Dermatitis subjects who take bleach baths two times per week for three months. The assumption was that this worked by reducing the S. aureus on the skin surface but by standard culture techniques there was no change in S. aureus colonization. Therefore, the mechanism by which these bleach baths improved the disease remains entirely unknown. This study will assess the effects bleach baths have on bacteria that can and cannot be cultured using new molecular biologic tools that have shown us that the skin is home to thousands of different microbial species. This bacterial ecosystem is called the microbiome. The investigators will also determine whether bleach baths affect skin barrier integrity and the cutaneous expression of lymphocyte-derived cytokines that are thought to cause the skin inflammation in subjects with Atopic Dermatitis. The investigators will also assess to what degree these baths improve disease severity and the symptoms of itch using validated scoring systems. This work will likely uncover new ideas about the pathogenesis of Atopic Dermatitis and may be the first step to developing new pro-microbial and antimicrobial therapeutics.

This study is designed to test the following hypotheses:

1. The chronic use of bleach baths will normalize skin barrier function in adult Atopic Dermatitis subjects as measured by physiological measures of barrier in vivo, and as assessed by ex vivo studies (measuring transepithelial electrical resistance (TEER) and permeability of the epidermis from skin biopsies). The investigators will evaluate whether any of the functional changes correlate with changes in expression of relevant tight and intercellular junction molecules at the messenger ribonucleic acid (mRNA) level.
2. Bleach baths will improve validated measures of pruritus (itch).
3. Bleach baths will diminish the local T-helper 2 (Th2) immune response measured from skin biopsy samples.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe Atopic dermatitis: Eczema Area and Severity Index (EASI) score ≥ 10.
* Skin culture positive for Staphylococcus aureus
* Must have active skin disease on the day of enrollment.

Exclusion Criteria:

* Unwillingness or inability to complete informed consent
* Lidocaine or Novocain allergy
* History of keloid formation
* Course of systemic antibiotics or antivirals within 2 weeks prior to enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-01; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Noninvasive barrier measurement called Transepidermal Water Loss (TEWL) done before and after repeated tape stripping | change from baseline after 12 weeks of bleach baths
  TEWL will be measured at 3 timepoints throughout the study.

SECONDARY OUTCOMES:
Itch - 5D pruritus scale | change from baseline after 12 weeks of bleach baths
  Change in self reported itch using a validated assessment tool.
Skin permeability | change from baseline after 12 weeks of bleach baths
  amount of fluorescent labeled molecule passage through the epithelial layer ex-vivo
Transepithelial electrical resistance | change from baseline after 12 weeks of bleach baths
  change of epithelium membrane potential and resistance in millivolts ex-vivo
Tissue expression of relevant inflammatory and epidermal barrier markers | change from baseline after 12 weeks of bleach baths
  Messenger ribonucleic acid (mRNA) expression of key inflammatory mediators and epidermal barrier proteins performed on the biopsy specimens
Skin bacterial diversity | change from baseline after 12 weeks of bleach baths
  Change in diversity of bacteria present in the skin

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Beck, MD, Principal Investigator — Department of Dermatology University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang JT, Abrams M, Tlougan B, Rademaker A, Paller AS. Treatment of Staphylococcus aureus colonization in atopic dermatitis decreases disease severity. Pediatrics. 2009 May;123(5):e808-14. doi: 10.1542/peds.2008-2217. PMID 19403473
- [Background] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Background] De Benedetto A, Rafaels NM, McGirt LY, Ivanov AI, Georas SN, Cheadle C, Berger AE, Zhang K, Vidyasagar S, Yoshida T, Boguniewicz M, Hata T, Schneider LC, Hanifin JM, Gallo RL, Novak N, Weidinger S, Beaty TH, Leung DY, Barnes KC, Beck LA. Tight junction defects in patients with atopic dermatitis. J Allergy Clin Immunol. 2011 Mar;127(3):773-86.e1-7. doi: 10.1016/j.jaci.2010.10.018. Epub 2010 Dec 15. PMID 21163515
- [Derived] Stolarczyk A, Perez-Nazario N, Knowlden SA, Chinchilli E, Grier A, Paller A, Gill SR, De Benedetto A, Yoshida T, Beck LA. Bleach baths enhance skin barrier, reduce itch but do not normalize skin dysbiosis in atopic dermatitis. Arch Dermatol Res. 2023 Dec;315(10):2883-2892. doi: 10.1007/s00403-023-02723-1. Epub 2023 Sep 27. PMID 37755506